CLINICAL TRIAL: NCT02987465
Title: An Observational, Open-label Pilot Study to Evaluate the Effect of Standard-of-care Erythropoiesis-stimulating Agents (Darbepoetin Alfa) on Forearm Blood Flow in Nondialysis-dependent Subjects With Anaemia Associated With Chronic Kidney Disease.
Brief Title: Evaluating the Effect of Standard-of-care Erythropoiesis-stimulating Agents on Forearm Blood Flow in Nondialysis-dependent Subjects With Anaemia Associated With Chronic Kidney Disease.
Acronym: OPERA-CKD
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician & Clinical Pharmacologist/Assoc Lecturer, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: OPERA-CKD (AO94224)
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Chronic Kidney Disease
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa; Acetylcholine; Norepinephrine; cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Some serum samples will be collected and stored for future analysis as part of the OPERA-CKD study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease patients: Up to 12 patients with anaemia associated with CKD.
  Interventions: Drug: Darbepoetin Alfa; Drug: Acetylcholine; Drug: Noradrenaline; Drug: BQ 123
- Healthy Volunteers: Up to 12 healthy subjects will be recruited such that age and gender are similar to the CKD patients. These subjects will be recruited as negative controls for a baseline assessment of healthy physiology. These subjects will not be treated with Darbepoetin.
  Interventions: Drug: Acetylcholine; Drug: Noradrenaline; Drug: BQ 123

INTERVENTIONS:
Drug: Darbepoetin Alfa — Darbepoetin is not a study drug and is prescribed as part of routine treatment of anaemia in CKD1. Darbepoetin is licensed for use for the treatment of anaemia in the context of CKD. It will be provided as part of the standard clinical care of the renal patients in this study. Healthy Volunteers will not be treated with Darbepoetin.
  Groups: Chronic Kidney Disease patients
Drug: Acetylcholine — Acetylcholine is being used as a challenge agent in this study and assesses NO-mediated vasodilation
Drug: Noradrenaline — Noradrenaline is being used as a challenge agent in this study and is an endogenous a1 adrenoceptor agonist
Drug: BQ 123 — BQ 123 is being used as a challenge agent in this study and is an (Endothelin A) ETA receptor agonist.

SUMMARY:
In people diagnosed with chronic kidney disease (CKD) anaemia is a common problem and is often treated with EPO (Erythropoietin). One form of EPO used is Darbepoetin (Aranesp®). EPO is safe to use but it has been associated with a rise in blood pressure (BP) in some individuals. The reasons for this are not clear. To try to explain this, this study will look at how EPO affects certain substances in the blood that influence how blood vessels contract and relax. This will be conducted by infusing small amounts of Acetylcholine, BQ123 and Noradrenaline into the arm vessels of volunteers using an established method called Forearm blood flow (plethysmography). Volunteers recruited for this study will include CKD patients undergoing therapy with Darbepoetin as part of their normal NHS care as well as healthy people not on treatment, who will act as controls. This is an observational pilot study of changes in physiology before and after Darbepoetin. It will provide valuable data for a later study comparing Darbepoetin to novel agents which work via different pathways to treat anaemia.

DETAILED DESCRIPTION:
This is a pilot proposal to understand the changes in physiology in patients undergoing scheduled therapy with Darbepoetin as part of their normal NHS care. It is therefore an observational pilot study of changes in physiology before and after Darbepoetin. Conventional erythropoiesis stimulating agents (ESAs) are widely used to improve haemoglobin production and reduce anaemia in subjects with chronic kidney disease (CKD). However, ESAs are associated with the development of hypertension and increased cardiovascular morbidity and mortality. A number of potential underlying pathophysiological mechanisms have been postulated, mostly concerning around altered sensitivity to, or circulating levels of, endogenous vasoactive mediators. However, the existing data are inconsistent. Hand et al. found that short-term therapy with recombinant erythropoietin was associated with a rise in blood pressure, and an increase in vasoconstrictor responsiveness to infused noradrenaline, but not to endothelin-1. Serum endothelin-1 levels were elevated compared to controls at baseline, but did not change after erythropoietin therapy. Other groups have reported that ESA administration increases plasma levels of endothelin-1, and that this is strongly correlated with the increase in mean arterial pressure (MAP). Human endothelial cells incubated in ESAs show decreased eNOS expression and endothelial nitric oxide (NO) production. Ex-vivo studies in resistance vessels of subjects with CKD found impaired endothelial function, as assessed by acetylcholine mediated vasodilatation, which was partially reversed by blockade of the endothelin receptor (ET-A). In vivo acute and chronic ESA administration also impairs endothelial function, which is often considered as a surrogate of nitric oxide bioavailability.

Recently, newer agents have been postulated as a novel alternative to ESAs for treating renal anaemia. However, cardiovascular effects are incompletely characterised. Studies elucidating the mechanisms for ESA induced vasoconstriction and possible effects that promote cardiovascular disease are necessary and it would be imperative to study whether the use of these novel agents avoids these effects, potentially making them a better alternative to ESAs.

This pilot study aims to determine the putative mechanisms which may be involved in the BP response to ESA use in patients with anaemia associated with CKD who are EPO naïve within the last 12 months. Information gained from this study will inform a larger clinical trial that is being planned. Healthy volunteers will be recruited to provide a baseline of normal responses to compare against.

ELIGIBILITY:
Inclusion Criteria CKD patients:

* Provided written informed consent to participate
* Be aged 18 years or over
* Clinically suitable for EPO (Darbepoetin) therapy as part of routine NHS standard of care for anaemia due to chronic kidney disease (CKD)
* No prior EPO treatment within the preceding 12 months
* Palpable brachial artery

Inclusion Criteria Healthy Volunteers:

* Provided written informed consent to participate
* Aged 18 years or over
* Blood pressure <140/90
* Normal haematology and renal function (defined as a normal creatinine and eGFR measured at any time in the last 6 months or at screening)
* Not on any regular prescribed medication
* Palpable brachial artery

Exclusion criteria CKD patients:

* Kidney transplant: Planned living-related kidney transplant within 26 weeks
* Patients on PDE5 inhibitors, alpha blockers, or nitrates (other than PRN GTN), unless they can be omitted until after the forearm study on the day of the visit
* MI or acute coronary syndrome in the preceding ≤ 4 weeks prior to screening
* Stroke or transient ischemic attack in the preceding ≤ 4 weeks prior to screening
* Known clinical diagnosis of Heart failure: NYHA Class III-IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Clinic Blood pressure: sustained BP > 170/100 mm Hg (on repeated measurements)
* Pregnancy - Non-sterilised, pre-menopausal women will undergo urinary beta-HCG testing at every visit and be given advice on contraceptive use in the PIS.
* Any other reason for exclusion from this study in the opinion of the Principal Investigator

Exclusion Criteria Healthy Volunteers:

* Any condition which, in the opinion of the investigator, precludes enrolment
* Undergoing investigation for any serious medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 12 patients with anaemia associated with chronic kidney disease (CKD).
  Up to 12 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Response to intra-arterial acetylcholine | CKD patients: Measured at baseline and at the end of the 6 week treatment period
  Change in forearm blood flow responses as measured by venous occlusion plethysmography, in response to intra-arterial acetylcholine

SECONDARY OUTCOMES:
Response to intra-arterial Noradrenaline | CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Change in forearm blood flow responses, as measured by venous occlusion plethysmography, in response to intra-arterial Noradrenaline
Response to intra-arterial BQ123 | CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Change in forearm blood flow responses as measured by venous occlusion plethysmography, in response to intra-arterial BQ123
Change in mean arterial blood pressure | CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Change in mean arterial blood pressure, systolic blood pressure and diastolic blood pressure post-Darbepoetin-Alfa over 6 weeks of treatment
Changes in Arterial stiffness | CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Changes in arterial stiffness post-darbepoetin-alfa
Correlations between individual challenge agent | CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Correlations between individual challenge agent forearm blood flow responses and change in blood pressure
Forearm blood flow responses to Acetylcholine, Noradrenaline and BQ123 in patients with CKD compared to healthy volunteers | Healthy Volunteers: Measured at baseline; CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Change in forearm blood flow responses to Acetylcholine, Noradrenaline and BQ123 in patients with anaemia associated with CKD at baseline compared to healthy volunteers
Responses to Acetylcholine, Noradrenaline and BQ123 in patients with CKD post-Darbepoetin compared to healthy volunteers | Healthy Volunteers: Measured at baseline; CKD patients: Measured at baseline before treatment with Darbepoetin and then at the end of the 6 week treatment period with Darbepoetin
  Change in forearm blood flow responses to Acetylcholine, Noradrenaline and BQ123 in patients with anaemia associated with CKD post-Darbepoetin compared to healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBCHB, MA, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided